CLINICAL TRIAL: NCT04764032
Title: Right Ventricular Dysfunction in Ventilated Patients With COVID-19
Acronym: COVID-RV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: Golden Jubilee National Hospital (Other Government); Robertson Centre for Biostatistics (Unknown)
Responsible Party: Principal Investigator, Dr Ben Shelley, Honorary Clinical Associate Professor, University of Glasgow
Other Study IDs: 20/COVID/17
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Right Ventricular Dysfunction; ARDS
Keywords: COVID-19; Right Ventricle; Echocardiography; ARDS
MeSH Terms: conditions — COVID-19; Ventricular Dysfunction, Right | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography will be undertaken by a range of appropriately competent practitioners including; intensive care clinicians, cardiologists and specialist echocardiographers. Imaging obtained will be in keeping with the protocol required for a Focused Intensive Care Echo (FICE) scan and should include ECG monitoring at all times. A focused dataset will be used to answer the primary outcome. If available and the echocardiographers competency and experience permit, further measures of RV function will be obtained at this time.

SUMMARY:
Using echocardiography to investigate the incidence of RV dysfunction in ventilated patients with COVID-19.

DETAILED DESCRIPTION:
INTRODUCTION Following the first reported cases in China, there has been a worldwide pandemic of a new virus commonly known as, Coronavirus. The virus causes a number of conditions including; cough, high temperature, painful muscles and breathing difficulties. The disease the virus causes is known as Coronavirus Disease 2019 (COVID-19). In the majority of cases these symptoms will get better without any treatment and without needing admission to hospital. In a small proportion of cases, the symptoms can be so bad that patients will need admission to hospital. Of the group admitted to hospital an even smaller group (approximately 5% of all confirmed coronavirus cases) will need treatment in an intensive care unit. This is often for severe breathing difficulties and sometimes requires the patient to be put on a breathing machine. The breathing machine is also known as a life support machine or ventilator and needing its support is known as 'ventilation' or 'being ventilated'.

In other conditions causing severe breathing difficulties requiring ventilation, pressure can be put on the right side of the heart ('the right heart [or right ventricle];' the part of the heart pumping blood to the lungs). This can cause the right heart to fail, struggling to pump blood forward and with a build-up of back pressure. This is also known as right heart (or ventricular) dysfunction. Patients needing ventilated, who develop problems with the right heart, are less likely to survive their intensive care stay. No scientists have examined whether patients with COVID-19, requiring ventilation, have problems with their right heart.

METHODS Using noninvasive ultrasound scans of the heart (echocardiography) the investigators will explore whether ventilated patients in intensive care have problems with their right heart. The investigators will also collect blood samples to look for damage to the heart during this time.

AIMS The aim of this study is to determine how many patients with COVID-19 needing ventilation have problems with the right heart. The investigators will explore if those patients with right heart problems are more likely to die by 30 days following their intensive care admission. By examining clinical data, the investigators will also look to see if any other conditions or treatments increase the risk of right heart problems. By identifying right heart problems in these patients, the investigators may be able to guide future studies to determine if any specific treatments targeted at protecting the right heart can improve outcomes in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Age > 16 years.
* Confirmed SARS-CoV-2 infection with severe acute respiratory failure requiring tracheal intubation and positive pressure ventilation in intensive care for more than 48 hours.

Exclusion Criteria:

* Pregnancy.
* Ongoing participation in any investigational research that may undermine the scientific basis of the study.
* Prior participation in the COVID-RV study.
* Ventilated for less than 48 hours prior to study recruitment.
* Those patients requiring extra-corporeal life support for respiratory or cardiovascular failure (veno-venous [VV] or veno-arterial [VA] extra-corporeal membrane oxygenation [ECMO]).
* Patient where end of life care has been instituted and they are not expected to survive for the next 24 hours.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring tracheal intubation and intermittent positive pressure ventilation for COVID-19 in Scottish intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
The prevalence of RV dysfunction in ventilated patients with COVID-19 | Any timepoint from eligibility (ventilation for more than 48 hours) to 14 days following tracheal intubation and positive pressure ventilation.
  RV dysfunction will be defined as Trans Thoracic Echo (TTE) evidence of RV dilatation along with the presence of septal flattening (in systole, diastole or both).
Association of RV dysfunction with 30-day mortality. | Up to 30-days following intubation and intermittent positive pressure ventilation

SECONDARY OUTCOMES:
Association of ARDS and RV dysfunction | At time of echocardiography
Association of micro/macro thrombi and RV dysfunction | At time of echocardiography
The association of direct myocardial injury and RV dysfunction | At time of echocardiography
The association of ventilation and RV dysfunction | At time of echocardiography
Association of ARDS and 30-day mortality | Up to 30-days following intubation and intermittent positive pressure ventilation
Association of micro/macro thrombi and 30-day mortality | Up to 30-days following intubation and intermittent positive pressure ventilation
Association of direct myocardial injury and 30-day mortality | Up to 30-days following intubation and intermittent positive pressure ventilation
Association of ventilation and 30-day mortality | Up to 30-days following intubation and intermittent positive pressure ventilation
The difference in NP levels between patients with, and patients without, RV dysfunction. | At time of echocardiography
The difference in hsTn between patients with, and patients without, RV dysfunction. | At time of echocardiography
Association between hsTn and 30-day mortality in patients with, and patients without, RV dysfunction | Up to 30-days following intubation and intermittent positive pressure ventilation
Association between NP levels and 30-day mortality in patients with, and patients without, RV dysfunction | Up to 30-days following intubation and intermittent positive pressure ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Ben Shelley, MD, Study Director — University of Glasgow
Locations (11):
- United Kingdom (11):
  - Aberdeen Royal Infirmary, Aberdeen
  - Univeristy Hospital, Ayr, Ayr
  - Golden Jubilee National Hospital, Clydebank
  - Dumfries and Galloway Royal Infirmary, Dumfries
  - University Hospital Hairmyres, East Kilbride
  - Queen Elizabeth University Hospital, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Raigmore Hospital, Inverness
  - University Hospital, Crosshouse, Kilmarnock
  - Royal Alexandra hospital, Paisley
  - University Hospital, Wishaw, Wishaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willder JM, McCall P, Messow CM, Gillies M, Berry C, Shelley B. Study protocol for COVID-RV: a multicentre prospective observational cohort study of right ventricular dysfunction in ventilated patients with COVID-19. BMJ Open. 2021 Jan 13;11(1):e042098. doi: 10.1136/bmjopen-2020-042098. PMID 33441361
- [Derived] McErlane J, McCall P, Willder J, Berry C, Shelley B; COVID-RV investigators. Right ventricular free wall longitudinal strain is independently associated with mortality in mechanically ventilated patients with COVID-19. Ann Intensive Care. 2022 Nov 12;12(1):104. doi: 10.1186/s13613-022-01077-7. PMID 36370220